CLINICAL TRIAL: NCT03930043
Title: A Metagenome-wide Association Study of Gut Microbiota in Gastrointestinal Non-Hodgkin's Lymphoma Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Deputy Director of Hematology Department, Ruijin Hospital
Other Study IDs: NHL-MGWAS
Record Dates: First submitted 2019-04-25; First posted 2019-04-29 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Gastrointestinal Lymphoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Health Control
  Interventions: Diagnostic Test: Metagenomic shotgun sequencing
- Non-gastrointestinal Lymphoma
  Interventions: Diagnostic Test: Metagenomic shotgun sequencing
- Gastric Lymphoma
  Interventions: Diagnostic Test: Metagenomic shotgun sequencing
- Intestinal Lymphoma
  Interventions: Diagnostic Test: Metagenomic shotgun sequencing

INTERVENTIONS:
Diagnostic Test: Metagenomic shotgun sequencing — preforming metagenomic shotgun sequencing on patients' or volunteers' feces specimen

SUMMARY:
This is a observational study on the fecal microbiota in primary/secondary gastrointestinal lymphoma patients.

DETAILED DESCRIPTION:
This observation study is aimed at investigating the gut microbiota alteration in gastrointestinal lymphoma (GIL) patients by performing metagenomic shotgun sequencing on GIL patients' fecal specimen. Before immuno-chemotherapy, the feces specimen of GIL would be collected and stored for further laboratory examination. This study would NOT alter the subsequential treatment of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal lymphoma with a clarified pathological diagnosis
* De novo gastrointestinal lymphoma patients who haven't received chemotherapy
* BMI in normal range

Exclusion Criteria:

* Antibiotics or probiotics application within a month
* Overweight (BMI≥25) or malnourished (BMI<18.5) patients
* Patients who have been accepted gastrointestinal fistulation
* Gastrointestinal patients with inflammatory bowel disease (IBD), colorectal carcinoma (CRC) or any other chronic intestinal disease
* Patients infected by HIV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The non-Hodgekin lymphoma patients with gastrointestinal involvement.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Metagenomic Linkage Groups (MLGs) | 2 years
  A serial of genes in a metagenome that is probably physically linked as a microbial unit.

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, MD. PhD., Study Chair — Ruijin Hospital
Locations (1):
- Shanghai Ruijin Hospital, Shanghai, Shanghai Municipality, China